CLINICAL TRIAL: NCT04572373
Title: Supplements SMOF in TPN for Liver Transplantation Recipients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201601322A3
Record Dates: First submitted 2020-09-14; First posted 2020-10-01 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Liver Transplantation; Total Parenteral Nutrition; End-stage Liver Disease
Keywords: Liver transplantation; SMOFlipid; fish oil
MeSH Terms: conditions — Hyperphagia; End Stage Liver Disease | interventions — SMOFlipid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SMOFlipid group: TPN and SMOFlipid support were indicated for patients who received NPO for more than 3 days, such as those with repeated laparotomy, staged biliary reconstruction, massive nasogastric (NG) drainage (>500 mL/day), ileus, diarrhoea, poor digestion (NG extraction >50 mL/time), and chylous ascites.
  Furthermore, SMOFlipid was discontinued when the platelet count decreased to 40,000/μL or less. In all cases, heparinisation was prescribed to maintain the aPTT level between 1.5 and 2 times the normal controlled level at least for 10-14 days, with daily blood examination conducted. Oral administration of dipyridamole (75 mg, QID) for 3 months was indicated for stimulation of antiplatelet activity when the platelet count increased to 40,000/μL or more.
  Interventions: Dietary Supplement: SMOFlipid
- non SMOFlipid group: On the basis of our experience in patient management at this institute, we allocated patients with a pretransplant platelet count less than 40,000/μL and those with a count more than 40,000/μL to the non-SMOFlipid group and the SMOFlipid group , respectively. Patients with well-tolerated oral intake and those in whom the TPN supplement was discontinued within 10 days were excluded from this study.

INTERVENTIONS:
Dietary Supplement: SMOFlipid
  Groups: SMOFlipid group

SUMMARY:
Liver transplantation (LT) is one of the widely recognised and leading treatments for end-stage liver disease. Nutrition impacts its success. Total parenteral nutrition (TPN) is usually prescribed for patients recommended prolonged fasting after LT. The supplement of SMOFlipid (soybean oil, MCT oil, olive oil, and fish oil) is easily metabolised to produce energy, and it possesses anti-inflammatory effects; however, SMOFlipid emulsion use raises concerns regarding coagulopathy after LT. This study investigated the postoperative correlation between SMOFlipid and coagulation in LT.

DETAILED DESCRIPTION:
Liver failure is characterised by the loss of liver function and is complicated with hepatic encephalopathy and coagulopathy. Liver transplantation (LT) is one of the widely recognised and leading treatments for end-stage liver disease. Malnutrition is one of the common manifestations of this critical condition and is also an independent predictor of mortality. Several studies have shown that malnutrition is a poor prognostic factor for LT, which indicates that nutritional support may reduce LT complications and improve survival.

Total parenteral nutrition (TPN) is usually prescribed for patients recommended prolonged fasting after LT. The supplement of SMOFlipid (soybean oil, MCT oil, olive oil, and fish oil) has the advantage of being easily metabolised to produce energy, and it has anti-inflammatory effects. The major therapeutic mechanism of fish oil is the attenuation of systematic inflammation, which may decrease the mortality risk in patients with severe injury and sepsis. SMOFlipid has been proven to be safe and well tolerated in a wide range of clinical conditions, and it is used as the standard lipid emulsion. Moreover, the short-term application of parenteral fish oil with soybean oil not only significantly reduces the parameters of liver damage in the postoperative period but also leads to a more balanced immune response, which may result in the faster resolution of inflammation and recovery. However, SMOFlipid emulsion use may be associated with coagulopathy after LT. Early studies have shown that the dietary intake of n-3 fatty acids, which is a component of fat, is associated with antithrombotic effects but increases the risk of bleeding. A detailed analysis is lacking, and these observations have yet to be proven; this concern persists. Hence, the investigators should pay attention to the bleeding tendency when using fish oil fat emulsion because it may aggravate the risk of bleeding. Therefore, the use of fish oil-containing fat emulsion and its related risks is a clinically important issue in early LT that should be investigated, because liver function is not restored immediately after transplantation, and there is a tendency of coagulopathy. Thus, classical haemostasis parameters such as activated partial thromboplastin time (aPTT) and platelet count are measured prior to surgery and before the start of TPN. However, many questions remain unanswered regarding nutritional assessment and support for these seriously ill, nutritionally, and metabolically complex patients. This study evaluated the effect of the SMOFlipid supplement in TPN in LT patients.

ELIGIBILITY:
Inclusion Criteria:

Adult (age > 18 years) LT recipients were enrolled

Exclusion Criteria:

1. Renal dysfunction (eGFR < 60 mL/min/1.73 m2)
2. Patients with well-tolerated oral intake and those in whom the TPN supplement was discontinued within 10 days were excluded from this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent LT at KCGMH between Jan 2012 and June 2015 were screened in this study. The medical records of patients were retrospectively reviewed to check if TPN was provided in the last 14 days in the peri-transplantation period. TPN and SMOFlipid support were indicated for patients who received NPO for more than 3 days, such as those with repeated laparotomy, staged biliary reconstruction, massive nasogastric (NG) drainage (>500 mL/day), ileus, diarrhoea, poor digestion (NG extraction >50 mL/time), and chylous ascites.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Patient demographics and clinical characteristics of SMOFlipid and non-SMOFlipid groups | 30 days
  Medical records including patient demographics, preoperative history, physical examination, clinical course, laboratory studies, aetiology of liver disease, severity of liver disease including Child-Pugh score and the Model for End-Stage Liver Disease (MELD) score, postoperative complications, and length of ICU and hospital stay were collected and reviewed.
Coagulopathy profile and nutrition profile in SMOF group and non-SMOFlipid groups | 30 days
  Medical records including laboratory studies (PT (sec), INR (sec), aPTT (sec), Platelet (103/uL), Albumin (g/dL), Cholesterol (mg/dL), Triglyceride (mg/dL))

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Che Lin, MD, Study Director — Department of Surgery, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Niaosong District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Koffron A, Stein JA. Liver transplantation: indications, pretransplant evaluation, surgery, and posttransplant complications. Med Clin North Am. 2008 Jul;92(4):861-88, ix. doi: 10.1016/j.mcna.2008.03.008. PMID 18570946
- [Result] Merli M, Giusto M, Giannelli V, Lucidi C, Riggio O. Nutritional status and liver transplantation. J Clin Exp Hepatol. 2011 Dec;1(3):190-8. doi: 10.1016/S0973-6883(11)60237-5. Epub 2012 Jan 2. PMID 25755385
- [Result] Xu J, Yunshi Z, Li R. Immunonutrition in surgical patients. Curr Drug Targets. 2009 Aug;10(8):771-7. doi: 10.2174/138945009788982432. PMID 19702523
- [Result] Kerwin AJ, Nussbaum MS. Adjuvant nutrition management of patients with liver failure, including transplant. Surg Clin North Am. 2011 Jun;91(3):565-78. doi: 10.1016/j.suc.2011.02.010. Epub 2011 Apr 29. PMID 21621696
- [Result] Henkel AS, Buchman AL. Nutritional support in patients with chronic liver disease. Nat Clin Pract Gastroenterol Hepatol. 2006 Apr;3(4):202-9. doi: 10.1038/ncpgasthep0443. PMID 16582962
- [Result] Wei C, Hua J, Bin C, Klassen K. Impact of lipid emulsion containing fish oil on outcomes of surgical patients: systematic review of randomized controlled trials from Europe and Asia. Nutrition. 2010 May;26(5):474-81. doi: 10.1016/j.nut.2009.09.011. Epub 2010 Jan 29. PMID 20116213
- [Result] Manzanares W, Langlois PL, Dhaliwal R, Lemieux M, Heyland DK. Intravenous fish oil lipid emulsions in critically ill patients: an updated systematic review and meta-analysis. Crit Care. 2015 Apr 16;19(1):167. doi: 10.1186/s13054-015-0888-7. PMID 25879776
- [Result] Klek S, Chambrier C, Singer P, Rubin M, Bowling T, Staun M, Joly F, Rasmussen H, Strauss BJ, Wanten G, Smith R, Abraham A, Szczepanek K, Shaffer J. Four-week parenteral nutrition using a third generation lipid emulsion (SMOFlipid)--a double-blind, randomised, multicentre study in adults. Clin Nutr. 2013 Apr;32(2):224-31. doi: 10.1016/j.clnu.2012.06.011. Epub 2012 Jul 12. PMID 22796064
- [Result] Nandivada P, Fell GL, Gura KM, Puder M. Lipid emulsions in the treatment and prevention of parenteral nutrition-associated liver disease in infants and children. Am J Clin Nutr. 2016 Feb;103(2):629S-34S. doi: 10.3945/ajcn.114.103986. Epub 2016 Jan 20. PMID 26791189
- [Result] Zhu XH, Wu YF, Qiu YD, Jiang CP, Ding YT. Liver-protecting effects of omega-3 fish oil lipid emulsion in liver transplantation. World J Gastroenterol. 2012 Nov 14;18(42):6141-7. doi: 10.3748/wjg.v18.i42.6141. PMID 23155344
- [Result] Hammad A, Kaido T, Aliyev V, Mandato C, Uemoto S. Nutritional Therapy in Liver Transplantation. Nutrients. 2017 Oct 16;9(10):1126. doi: 10.3390/nu9101126. PMID 29035319
- [Result] Knapp HR. Dietary fatty acids in human thrombosis and hemostasis. Am J Clin Nutr. 1997 May;65(5 Suppl):1687S-1698S. doi: 10.1093/ajcn/65.5.1687S. PMID 9129511
- [Result] Heller AR, Fischer S, Rossel T, Geiger S, Siegert G, Ragaller M, Zimmermann T, Koch T. Impact of n-3 fatty acid supplemented parenteral nutrition on haemostasis patterns after major abdominal surgery. Br J Nutr. 2002 Jan;87 Suppl 1:S95-101. doi: 10.1079/bjn2001462. PMID 11895160
- [Result] Mateu de Antonio J, Florit-Sureda M. Effects unrelated to anti-inflammation of lipid emulsions containing fish oil in parenteral nutrition for adult patients. Nutr Hosp. 2017 Feb 1;34(1):193-203. doi: 10.20960/nh.882. PMID 28244792
- [Result] Starzl TE, Iwatsuki S, Esquivel CO, Todo S, Kam I, Lynch S, Gordon RD, Shaw BW Jr. Refinements in the surgical technique of liver transplantation. Semin Liver Dis. 1985 Nov;5(4):349-56. doi: 10.1055/s-2008-1040632. No abstract available. PMID 3909429
- [Result] Grewal HP, Shokouh-Amiri MH, Vera S, Stratta R, Bagous W, Gaber AO. Surgical technique for right lobe adult living donor liver transplantation without venovenous bypass or portocaval shunting and with duct-to-duct biliary reconstruction. Ann Surg. 2001 Apr;233(4):502-8. doi: 10.1097/00000658-200104000-00004. PMID 11303131
- [Result] Tanaka K, Uemoto S, Tokunaga Y, Fujita S, Sano K, Nishizawa T, Sawada H, Shirahase I, Kim HJ, Yamaoka Y, et al. Surgical techniques and innovations in living related liver transplantation. Ann Surg. 1993 Jan;217(1):82-91. doi: 10.1097/00000658-199301000-00014. PMID 8424706
- [Result] Inomata Y, Uemoto S, Asonuma K, Egawa H. Right lobe graft in living donor liver transplantation. Transplantation. 2000 Jan 27;69(2):258-64. doi: 10.1097/00007890-200001270-00011. PMID 10670636
- [Result] Stephenson GR, Moretti EW, El-Moalem H, Clavien PA, Tuttle-Newhall JE. Malnutrition in liver transplant patients: preoperative subjective global assessment is predictive of outcome after liver transplantation. Transplantation. 2001 Aug 27;72(4):666-70. doi: 10.1097/00007890-200108270-00018. PMID 11544428
- [Result] Wichmann MW, Thul P, Czarnetzki HD, Morlion BJ, Kemen M, Jauch KW. Evaluation of clinical safety and beneficial effects of a fish oil containing lipid emulsion (Lipoplus, MLF541): data from a prospective, randomized, multicenter trial. Crit Care Med. 2007 Mar;35(3):700-6. doi: 10.1097/01.CCM.0000257465.60287.AC. PMID 17261965
- [Result] Merli M, Giusto M, Gentili F, Novelli G, Ferretti G, Riggio O, Corradini SG, Siciliano M, Farcomeni A, Attili AF, Berloco P, Rossi M. Nutritional status: its influence on the outcome of patients undergoing liver transplantation. Liver Int. 2010 Feb;30(2):208-14. doi: 10.1111/j.1478-3231.2009.02135.x. Epub 2009 Oct 14. PMID 19840246
- [Result] Sukhotnik I, Shany A, Bashenko Y, Hayari L, Chemodanov E, Mogilner J, Coran AG, Shaoul R. Parenteral but not enteral omega-3 fatty acids (Omegaven) modulate intestinal regrowth after massive small bowel resection in rats. JPEN J Parenter Enteral Nutr. 2010 Sep-Oct;34(5):503-12. doi: 10.1177/0148607110362586. PMID 20852178
- [Result] Barbosa VM, Miles EA, Calhau C, Lafuente E, Calder PC. Effects of a fish oil containing lipid emulsion on plasma phospholipid fatty acids, inflammatory markers, and clinical outcomes in septic patients: a randomized, controlled clinical trial. Crit Care. 2010;14(1):R5. doi: 10.1186/cc8844. Epub 2010 Jan 19. PMID 20085628